CLINICAL TRIAL: NCT05956301
Title: Effects of Different Ventilatory Strategy During Bronchoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Liya Lu, associate chief physician, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230618
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Bronchoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Conventional Oxygen Therapy
  Interventions: Device: Conventional Oxygen Therapy
- Group II (Experimental): High-flow nasal oxygen
  Interventions: Device: High-flow nasal oxygen
- Group III (Experimental): Supraglottic jet oxygenation and ventilation
  Interventions: Device: Supraglottic jet oxygenation and ventilation

INTERVENTIONS:
Device: Conventional Oxygen Therapy — Conventional Oxygen Therapy will be administered through Nasal catheter
  Arms: Group I
Device: High-flow nasal oxygen — High Flow Nasal Cannula will be administered
  Arms: Group II
Device: Supraglottic jet oxygenation and ventilation — Nasal jet tube will be administered
  Arms: Group III

SUMMARY:
The execution of diagnostic-therapeutic investigations by bronchial endoscopy can expose the patient to hypoxemia. For this reason, oxygen therapy is administered at low or high flows during the course of bronchoscopic procedures.

Our study aim was to evaluate the efficacy and complications of High-flow nasal oxygen (HFNO) via Supraglottic jet oxygenation and ventilation (SJOV)during flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* need for bronchial endoscopy

Exclusion Criteria:

* life-threatening cardiac aritmia or acute miocardical infarction within 6 weeks need for invasive or non invasive ventilation presence of pneumothorax or pulmonary enphisema or bullae recent (within 1 week) thoracic surgery presence of chest burns presence of tracheostomy pregnancy nasal or nasopharyngeal diseases dementia lack of consent or its withdrawal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the intraoperative oxygenation. | During bronchoscopy, an average of 0.5 hour.
  The study will monitor the SpO2， heart rate(HR) and mean arterial pressure (MAP) during the procedure.

SECONDARY OUTCOMES:
Arterial blood gases | At end of of bronchoscopy,an average of 0.5 hour after bronchoscope insertion.
  Arterial blood gas analysis will be monitored at end of of procedure.
Assess the regional ventilation distribution by Electrical impedance tomography . | During bronchoscopy, an average of 0.5 hour.
  Measurements will be done after bronchoscope insertion and at the end of the procedure.